CLINICAL TRIAL: NCT06756880
Title: The Role of Preoperative Pulmonary Function Tests in Predicting Postoperative Intensive Care Need in Adolescent Idiopathic Scoliosis Surgery: A Retrospective Cohort Study
Brief Title: Prognostic Significance of Pulmonary Function Tests in Adolescent İdiopathic Scoliosis Surgery
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Gökhan Erdem, Anesthesiology and Reanimation specialist doctor, Ankara City Hospital Bilkent
Other Study IDs: AIS
Record Dates: First submitted 2024-12-24; First posted 2025-01-03 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Anesthesia; Pulmonary Function Test, Preoperative; Adolescent Idiopathic Scoliosis
Keywords: Adolescent Idiopathic Scoliosis; Preoperative Pulmonary Function Test
MeSH Terms: interventions — Respiratory Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- normal risk: z score is greater than -1.645
  Interventions: Diagnostic Test: Pulmonary function test
- Low risk: z score between -1.645 and -2.5
  Interventions: Diagnostic Test: Pulmonary function test
- Medium risk: z score between -2.5 and -4.0
  Interventions: Diagnostic Test: Pulmonary function test
- High risk: z score of less than -4.0
  Interventions: Diagnostic Test: Pulmonary function test

INTERVENTIONS:
Diagnostic Test: Pulmonary function test — Pulmonary function test results performed closest to the date of surgery and considered successful according to American Thoracic Society standards

SUMMARY:
Adolescent idiopathic scoliosis (AIS) is a three-dimensional structural deformity of the spine, the etiology of which is not clearly known, and can be seen from the age of 10 until the skeletal system matures. The Scoliosis Research Society (SRS) defines AIS as vertebral rotation and a Cobb angle of 10° or greater. Its incidence varies between 0.47% and 5.2%. It is more common in women than in men. In patients with a Cobb angle greater than 40° or who are not yet bone-mature and who are continuously progressing, surgical intervention is often performed with posterior spinal fusion. Scoliosis negatively affects not only the appearance of patients but also their lung functions through differentiation in thoracic morphology and progression of spinal curvature. The severity of this restrictive pattern in lung functions can be assessed with pulmonary function tests (PFT). However, this test requires patient cooperation and is particularly difficult to perform in patients with cognitive dysfunction. Despite studies recommending the use of pulmonary function tests in preoperative risk assessment, the literature shows inconsistency in predicting the need for postoperative intubation and mechanical ventilation.

In this study, the effect of preoperative pulmonary function tests (PFT) performed before AIS surgery on the need for intensive care admission will be evaluated. In addition, the potential relationships between PFT results and intraoperative and postoperative blood transfusion needs, postoperative intubation needs, hospital stay, mortality status, inotropic support needs, Cobb angle, scoliosis location, and the number of affected vertebrae will be investigated.

DETAILED DESCRIPTION:
After local ethics committee approval, patients' age, gender, weight, American Society of Anesthesiologists (ASA) physical status, additional diseases, localization of scoliosis, number of vertebrae affected, Cobb angle and presence of chronic lung disease will be recorded within the scope of demographic data.

Cobb angle or lateral spinal curvature will be measured and recorded on the spine radiograph closest to the date of surgery. In terms of preoperative respiratory function tests, the results performed closest to the date of surgery and accepted as successful according to American Thoracic Society standards will be analyzed. In this context, forced vital capacity (FVC) percentage of normal, forced expiratory volume in 1 second (FEV1) percentage of normal, and FEV1/FVC ratios will be recorded. In the presence of an obstructive or restrictive pattern, FEV1/FVC or FVC Z-scores will be examined and evaluated as normal, mild, moderate or severe in accordance with European Respiratory Society/American Thoracic Society (ERS/ATS) guidelines. The Z-score shows how much the individual's measured value deviates from the reference population determined according to factors such as ethnicity, gender, age, and height. A z-score greater than -1.645 is considered normal, a z-score between -1.645 and -2.5 is considered mild, a z-score between -2.5 and -4.0 is considered moderate, and a z-score below -4.0 is considered severe.

The recorded data will be evaluated by considering the need for intensive care admission, need for intraoperative and postoperative blood transfusion, need for postoperative intubation, length of hospital stay, mortality status, need for inotropic support, Cobb angle, location of scoliosis and number of affected vertebrae. Postoperative intubation status will be defined as patients brought to the ICU without extubation or re-intubated within 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Age range 10-18
* Patients who underwent posterior spinal fusion surgery for Adolescent Idiopathic Scoliosis under general anesthesia

Exclusion Criteria:

* Body mass index >35 kg/m²
* ASA (American Society of Anesthesiologists) score of 4 and above
* Patients who have undergone revision surgery
* Patients with mental retardation
* Need for Bilevel Positive Airway Pressure (BPAP) before surgery
* Patients who could not successfully complete preoperative respiratory function tests
* Preoperative tracheostomy presence
* Patients with vertebral anomaly due to a secondary reason
* Patients with a diagnosed syndrome

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients between the ages of 10-18 who underwent posterior spinal fusion surgery under general anesthesia due to Adolescent Idiopathic Scoliosis (AIS) will be included in the study. Exclusion criteria were determined as ASA (American Society of Anesthesiologists) score of 4 and above, body mass index >35 kg/m², mental retardation, Need for Bilevel Positive Airway Pressure (BPAP) before surgery, patients who could not successfully complete preoperative respiratory function tests, presence of tracheostomy and revision surgeries.
Sampling Method: Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Need for intensive care admission | 2019 - 2024
  The primary outcome of the study was to evaluate the effect of preoperative lung function tests performed before adolescent idiopathic scoliosis surgery on the need for postoperative intensive care admission.

SECONDARY OUTCOMES:
Hospital stay | 2019 - 2024
  Investigation of the potential relationship between pulmonary function test results and hospital stay
Need for blood transfusion | 2019 - 2024
  Investigation of the potential relationship between pulmonary function test results and need for blood transfusion
Mortality status | 2019 - 2024
  Investigation of the potential relationship between pulmonary function test results and mortality status
İnotropic support requirement | 2019 - 2024
  Investigation of the potential relationship between pulmonary function test results and inotropic support requirement
Cobb angle | 2019 - 2024
  Investigation of the potential relationship between pulmonary function test results and cobb angle
Location of scoliosis and number of affected vertebrae | 2019 - 2024
  Investigation of the potential relationship between pulmonary function test results and location of scoliosis and number of affected vertebrae
Need for postoperative intubation | 2019 - 2024
  Investigation of the possible relationship between lung function test results and the need for postoperative intubation Postoperative intubation status was defined as patients brought to the ICU without extubation or reintubated within 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No